CLINICAL TRIAL: NCT04776408
Title: Potential for Inhaled Nitric Oxide and Ventilation-Perfusion Mismatch by Electrical Impedance Tomography in the Acute Respiratory Distress Syndrome Patients With Lung Recruitment
Brief Title: Potential for Inhaled Nitric Oxide and Ventilation-Perfusion Mismatch by Electrical Impedance Tomography in the ARDS Patients With Lung Recruitment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109200-F
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-02

CONDITIONS: Nitric Oxide; Acute Respiratory Distress Syndrome
Keywords: Electrical Impedance Tomography; Acute Respiratory Distress Syndrome; Inhaled Nitric Oxide; Ventilation-Perfusion mismatch; Lung recruitment
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Moderate to severe ARDS patient on mechanical ventilation in Far Eastern Memorial Hospital MICU
Who Masked: Participant
Masking Description: During this period, all patients were total sedation using continuous infusion, to prevent any spontaneous breathing .All patients were ventilated using a ventilator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group_Use Lung recruitment (Active Comparator): Use the Lung recruitment,
  Interventions: Device: Lung recruitment
- Study group_Use Lung recruitment combined inhaled Nitric oxide (Experimental): Use the Lung recruitment combined inhaled Nitric oxide,
  Interventions: Device: Lung recruitment combined inhaled Nitric oxide

INTERVENTIONS:
Device: Lung recruitment combined inhaled Nitric oxide — Ventilator combined inhaled Nitric oxide and Electrical Impedance Tomography monitor the V/Q mismatch
  Arms: Study group_Use Lung recruitment combined inhaled Nitric oxide
Device: Lung recruitment — Ventilator and Electrical Impedance Tomography monitor the V/Q mismatch
  Arms: Control group_Use Lung recruitment

SUMMARY:
In the recent years, the treatment of Acute Respiratory Distress Syndrome has been proved that lung recruitment re-opens the non-ventilated alveolar to improve ventilation, and inhaled Nitric Oxide dilates non-perfused pulmonary vascular to improve perfusion. Both of these could improve ventilation-perfusion mismatch to enhance oxygenation. However, Ventilation-Perfusion mismatch is devided into ventilated nonperfused lung units(dead space) or perfused nonventilated units(shunt). No published study has evaluated the availability of lung recruitment combined with inhaled Nitric oxide in patients with ARDS.

The aims of our study are to measure dead space or shunt fraction before and after inhaled Nitric Oxide in moderate to severe Acute Respiratory Distress Syndrome patients indicated Nitric oxide in FEMH MICU on 2021/01-2022/12, injected a bolus of 10mL of 3% NaCl solution via the central venous catheter with two-step recruitment maneuver by Electrical Impedance Tomography, which monitors ventilation-perfusion mismatch to evaluate whether the patient has potential to improve V/Q mismatch by Nitric oxide.

DETAILED DESCRIPTION:
Normally, pulmonary arteries in areas of alveolar hypoxia will constrict as a physiologic response to preserve ventilation/perfusion (V¬/Q¬) matching. However, in ARDS, this normal vasoconstrictive response is impaired. Because the body is unable to shunt blood away from the diseased alveoli, these nonaerated alveoli receive excessive blood flow, which contributes to severe V¬/Q¬ mismatching and an intrapulmonary right-to-left shunting of blood flow, which causes hypoxemia.

In the recent years, the treatment of Acute Respiratory Distress Syndrome has been proved that lung recruitment re-opens the non-ventilated alveolar to improve ventilation, and inhaled Nitric Oxide dilates non-perfused pulmonary vascular to improve perfusion. Both of these could improve ventilation-perfusion mismatch to enhance oxygenation. However, Ventilation-Perfusion mismatch is devided into ventilated nonperfused lung units(dead space) or perfused nonventilated units(shunt). No published study has evaluated the availability of lung recruitment combined with inhaled Nitric oxide in patients with ARDS.

The aims of our study are to measure dead space or shunt fraction before and after inhaled Nitric Oxide in moderate to severe Acute Respiratory Distress Syndrome patients indicated Nitric oxide in FEMH MICU on 2021/01-2022/12, injected a bolus of 10mL of 3% NaCl solution via the central venous catheter with two-step recruitment maneuver by Electrical Impedance Tomography, which monitors ventilation-perfusion mismatch to evaluate whether the patient has potential to improve V/Q mismatch by Nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS patient on mechanical ventilation in MICU. (P/F≦ 200 with PEEP ≥ 5cmH20) (PEEP greater than or equal to 5 cm H2O and Berlin criteria for ARDS)

Exclusion Criteria:

* Hemodynamic instability or severe COPD, pulmonary embolism
* Acute brain injury, seizure attack, AMI, AIDS, severe arrhythmia
* On pacemaker
* Pregnant
* Thoracic trauma or burn injury
* Pneumothorax

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
V/Q mismatch | 15 minutes
  Compare the V/Q mismatch between two groups

SECONDARY OUTCOMES:
PaO2/FiO2 ratio improvement rate | 15 minutes
  Oxygention improve rate

CONTACTS AND LOCATIONS:
Overall Officials: Hou T Chang, Doctor, Study Director — Far Eastern Memorial Hospital; Ping H Wang, Bachelor, Study Director — Far Eastern Memorial Hospital; Mei Y Chang, Master, Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Banqiao Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
Still in the research phase.May be consider later

REFERENCES:
- [Background] Bluth T, Kiss T, Kircher M, Braune A, Bozsak C, Huhle R, Scharffenberg M, Herzog M, Roegner J, Herzog P, Vivona L, Millone M, Dossel O, Andreeff M, Koch T, Kotzerke J, Stender B, Gama de Abreu M. Measurement of relative lung perfusion with electrical impedance and positron emission tomography: an experimental comparative study in pigs. Br J Anaesth. 2019 Aug;123(2):246-254. doi: 10.1016/j.bja.2019.04.056. Epub 2019 May 31. PMID 31160064
- [Background] Mauri T, Spinelli E, Scotti E, Colussi G, Basile MC, Crotti S, Tubiolo D, Tagliabue P, Zanella A, Grasselli G, Pesenti A. Potential for Lung Recruitment and Ventilation-Perfusion Mismatch in Patients With the Acute Respiratory Distress Syndrome From Coronavirus Disease 2019. Crit Care Med. 2020 Aug;48(8):1129-1134. doi: 10.1097/CCM.0000000000004386. PMID 32697482
- See also: Measurement of relative lung perfusion with electrical impedance and positron emission tomography: an experimental comparative study in pigs — https://pubmed.ncbi.nlm.nih.gov/31160064/
- See also: Potential for Lung Recruitment and Ventilation-Perfusion Mismatch in Patients With the Acute Respiratory Distress Syndrome From Coronavirus Disease 2019 — https://pubmed.ncbi.nlm.nih.gov/32697482/